CLINICAL TRIAL: NCT06558201
Title: Open Label Extension Study of NCT06221852 of the Ketogenic Diet in Participants With First Episode Bipolar Disorder.
Brief Title: Open Label Extension Study of NCT06221852
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Baszucki Family Foundation (Unknown)
Responsible Party: Principal Investigator, Virginie-Anne Chouinard, MD, Principal Investigator, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P002849-2
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Bipolar I Disorder; Schizoaffective Disorder; Psychosis
Keywords: First episode psychosis; Ketogenic diet; Keto; Brain energy metabolism; Insulin resistance; Schizoaffective disorder; Bipolar disorder; Magnetic resonance spectroscopy (MRS); Redox; Creatine kinase
MeSH Terms: conditions — Psychotic Disorders; Insulin Resistance; Bipolar Disorder | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: All participants will have completed the 12-week randomized controlled trial (NCT06221852), and will follow the ketogenic diet in this open label extension.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic diet (Experimental): Participants will be asked to follow the ketogenic diet (KD) for 12 weeks in addition to any ongoing medications (e.g., mood stabilizers and/or second-generation antipsychotics). Participants will receive diet counseling from a registered dietitian. Participants will be asked to monitor and report their blood ketone and glucose levels each day via a finger-prick device provided by the study team.
  Interventions: Other: Ketogenic diet

INTERVENTIONS:
Other: Ketogenic diet — The ketogenic diet (KD) is a normo-caloric diet composed of high-fat, low carbohydrate, and adequate protein intake. The KD will consist of 3 meals a day plus snacks, targeting 75-80% fat, 13-18% protein, 7% carbohydrates.
  Other Names: Keto diet

SUMMARY:
This is a 12-week open-label extension study for participants completing study NCT06221852.

DETAILED DESCRIPTION:
In this 12-week single arm open label extension study of NCT06221852, the investigators aim to assess the longer term efficacy, safety and tolerability of the ketogenic diet in participants completing the randomized study phase of NCT06221852. Investigators will assess longer term effects on energy metabolism, insulin resistance and psychiatric symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Participants who met original entry criteria in, and completed, the randomized 12-week study of NCT06221852.

Exclusion Criteria:

-No longer meeting original entry criteria from the randomized 12-week study of NCT06221852.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in brain redox nicotinamide adenine dinucleotide metabolites ratio (NAD+/NADH) | 24 weeks
  Change from baseline to week 24 in NAD+/NADH as measured by in vivo phosphorus magnetic resonance spectroscopy (31P-MRS).
Change in brain creatine kinase forward reaction rate (kf) | 24 weeks
  Change from baseline to week 24 in creatine kinase forward reaction rate (kf) as measured by 31P magnetization transfer (MT) MRS.
Change in insulin resistance | 24 weeks
  Change from baseline to week 24 of insulin resistance measured using the homeostatic model assessment of insulin resistance (HOMA-IR) using fasting blood glucose and insulin levels.
Change in psychotic symptoms | 24 weeks
  Change from baseline to week 24 in Positive and Negative Syndrome Scale (PANSS) total score. Scores range from 30-210; a higher score indicates a higher level of psychotic symptoms.
Change in depressive symptoms | 24 weeks
  Change from baseline to week 24 in Hamilton Rating Scale for Depression (HAM-D) total score. Scores range from 0-52; a higher score indicates a higher level of depression.
Change in mania symptoms | 24 weeks
  Change from baseline to week 24 in Young Mania Rating Scale (YMRS) total score. Scores range from 0-60. A higher score indicates a more severe illness.
Change in Clinical Global Impression (CGI) Scale | 24 weeks
  Change from baseline to week 24 in Clinical Global Impression (CGI) Scale. Scores range from 1-7; a higher score indicates higher severity of illness.

SECONDARY OUTCOMES:
Change in body weight | 24 weeks
  Change from baseline to week 24 in participant body weight in kilograms, as measured using a standing scale.
Change in glycated hemoglobin (Hemoglobin A1c) level | 24 weeks
  Change from baseline to week 24 in fasting Hemoglobin A1c level.
Change in triglyceride levels | 24 weeks
  Change from baseline to week 24 in fasting triglyceride levels.
Change in low-density lipoprotein (LDL) levels | 24 weeks
  Change from baseline to week 24 in fasting LDL levels
Change in high-density lipoprotein (HDL) levels | 24 weeks
  Change from baseline to week 24 in fasting HDL levels
Change in high-sensitivity C-reactive protein (hs-CRP) levels | 24 weeks
  Change from baseline to week 24 in fasting hs-CRP levels.
Change in brain gamma-aminobutyric acid (GABA) concentration | 24 weeks
  Change from baseline to week 24 in GABA concentration measured by proton magnetic resonance spectroscopy.
Change in brain glutamate metabolite concentration | 24 weeks
  Change from baseline to week 24 in glutamate metabolite concentration measured by proton magnetic resonance spectroscopy.
Change in brain glutathione (GSH) | 24 weeks
  Change from baseline to week 24 in brain GSH measured by proton magnetic resonance spectroscopy.
Change in brain Phosphocreatine (PCr) | 24 weeks
  Changes from baseline to week 24 in PCr concentration as measured by in vivo 31P-MRS.
Change in brain pH | 24 weeks
  Change from baseline to week 24 in pH as measured by in vivo 31P MRS
Change in brain inorganic phosphate concentration | 24 weeks
  Change from baseline to week 24 in inorganic phosphate (Pi) concentration as measured by in vivo 31P MRS.
Change in adverse events | 24 weeks
  Change from baseline to week 24 in adverse events.
Change in anxiety symptoms | 24 weeks
  Change from baseline to week 24 from baseline to week 12 in Hamilton Anxiety Rating Scale (HAM-A) total score. Scores range from 0 - 56; a higher score indicates a higher level of anxiety.
Change in stress symptoms | 24 weeks
  Change from baseline to week 24 in Depression Anxiety Stress Scales (DASS-42) Stress Subscale score. Scores range from 0-42; a higher score indicates a higher level of stress.
Change in cognitive performance | 24 weeks
  Change from baseline to week 24 in Matrics Consensus Cognitive Battery (MCCB) Total Score. Scores range from 0.00% - 100.00%; a higher score indicates higher cognition.
Change in Global Functioning Scale (GFS) - Social and Role total score | 24 weeks
  Change from baseline to week 24 in Global Functioning Scale (GFS) - Social and Role total score. Scores range from 6-60; a lower score indicates worse social and role functioning.
Change in blood NAD/NADH+ ratio | 24 weeks
  Change from baseline to week 24 in blood NAD/NADH+ ratio.
Change in blood GSH/GSSH ratio | 24 weeks
  Change from baseline to week 24 in blood GSH/GSSH ratio.
Change in growth differentiation factor 15 (GDF15) | 24 weeks
  Change from baseline to week 24 in blood and saliva GDF15 levels.
Change in cell-free mitochondrial DNA (cf-mtDNA) | 24 weeks
  Change from baseline to week 24 in blood and saliva cf-mtDNA levels.

OTHER OUTCOMES:
Change in World Health Organization Disability Assessment Schedule (WHODAS) score | 24 weeks
  Change from baseline to week 24 in World Health Organization Disability Assessment Schedule (WHODAS) scale. Scores range from 0-144. A higher score indicates greater dysfunction and disability in major life domains.
Change in World Health Organization Quality of Life (WHOQOL) score | 24 weeks
  Change from baseline to week 24 in World Health Organization Quality of Life (WHOQOL) scale. Scores range from 1-130. A lower score indicates lower perceived quality of life.
Change in Extrapyramidal Symptom Rating Scale (ESRS) total score | 24 weeks
  Change from baseline to week 24 in Extrapyramidal Symptom Rating Scale (ESRS) total score. Scores range from 0-102; a higher score indicates more severe symptoms.
Change in Pittsburgh Sleep Quality Index (PSQI) total score | 24 weeks
  Change from baseline to week 24 in Pittsburgh Sleep Quality Index (PSQI) total score. Scores range from 0-21; a higher score indicates worse sleep quality.
Change in resting-state fMRI | 24 weeks
  Change within network positive correlations and between network negative correlations from baseline to week 24.
Change in gray matter volume | 24 weeks
  Change in the gray matter volumes (cubic millimeters) of the frontal, parietal and temporal lobes as defined by Freesurfer's Desikan-Killiany Brain Atlas from baseline to week 24.
Change in cortical surface area | 24 weeks
  Change in the cortical surface area (millimeters squared) of the frontal, parietal and temporal lobes as defined by Freesurfer's Desikan-Killiany Brain Atlas from baseline to week 24.
Change in white matter fractional anisotropy (FA) | 24 weeks
  Change in fractional anisotropy (FA), a scalar measure of diffusivity, of water in the brain assessed by DTI at 3T from baseline to week 24. FA values range from 0 (isotropic, meaning diffusion is equally restricted in 3D space) to 1 (anisotrophic, meaning that diffusion is completely restricted to a single direction).

CONTACTS AND LOCATIONS:
Overall Officials: Virginie-Anne Chouinard, MD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States